CLINICAL TRIAL: NCT04197960
Title: A Prospective Multicenter Study to Compare the Therapeutic Outcomes of Microwave Ablation With Surgical Resection for Micropapillary Thyroid Carcinoma
Brief Title: Microwave Ablation and Surgical Resection for Micropapillary Thyroid Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Professor, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 301jrcsk-lp
Record Dates: First submitted 2019-12-04; First posted 2019-12-13 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2024-12

CONDITIONS: Papillary Thyroid Carcinoma
Keywords: Papillary Thyroid Carcinoma; Microwave ablation; Surgical resection
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- microwave ablation (Experimental): ablate all tumors including at least 2mm safe margin except for tumors adjacent to thyroid capsule.
  Interventions: Procedure: Microwave ablation
- surgical resection (Active Comparator): thyroid lobectomy, total thyroidectomy, central lymph node dissection
  Interventions: Procedure: Surgical resection

INTERVENTIONS:
Procedure: Microwave ablation — Use thermal energy to destroy tumor
  Arms: microwave ablation
Procedure: Surgical resection — Resect tumors
  Arms: surgical resection

SUMMARY:
The study aimed to compare the efficacy and safety of papillary thyroid microcarcinoma (PTMC) treated with microwave ablation(MWA) and surgery resection (SR), and to explore the tumor characteristics suitable for each treatment methods (such as with and without capsular invasion). The investigators organized 18 hospitals to participate in this multicenter study. Patients meeting following indications will be included in this study: 1. Biopsy pathology proved PTMC, but not high-risk subtype; 2. solitary mPTC, without US-detected gross extrathyroid extension; 3. no evidence of metastasis; 4 willing to participate in this study and perform regular follow-up. Patients themselves decide to receive MWA or SR for mPTC after medical consultation. Baseline characteristic including age, gender, thyroid function et al. will be collected. The treatment protocols of MWA and SR were according to the Chinese and international guidelines. The primary outcomes were the disease progression, including local tumor recurrence, lymph node metastasis, and distant metastasis. The secondary outcomes include thyroid function, complication rate, blood loss et al. Investigators will follow up enrolled patients and collect and upload data according to the trial. Treatment outcomes of tumor with and without US-detected capsular invasion was analyzes as subgroups.

DETAILED DESCRIPTION:
The treatment protocols of MWA and SR were according to the Chinese and international guidelines. MWA need to ablate all tumors including at least 2mm safe margin except for tumors adjacent to thyroid capsule. SR basic protocol is lobectomy. All patients need to receive levothyroxine therapy to keep TSH lower than 0.5 mU/L. Patients in both groups underwent regular medical imaging and laboratory tests 1 month, 3-month, 6-month, 12-month, 18-month, 24-month and 36-month after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy pathology proved micropapillary thyroid carcinoma(mPTC), but not high-risk subtype
* Solitary mPTC, without US-detected gross extrathyroid extension
* No evidence of metastasis
* Willing to participate in this study and perform regular follow-up

Exclusion Criteria:

* Severe blood coagulation dysfunction (platelet count < 50x109/L cells or INR>1.5)
* Acute or severe chronic renal failure, pulmonary insufficiency or heart dysfunction
* Poor control of blood pressure(systolic pressure≥150mmHg or diastolic pressure≥95mmHg)
* Poor control of blood glucose(fasting glucose>10mmol/L)
* The opposite vocal cords dysfunction
* Diagnosed with other malignant tumors
* Pregnant and lactating women
* Other conditions that investigator believe are not appropriate to be enrolled

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 973 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
local tumor progression | 2-year
  the number of patients with tumor progression around the treated area
lymph node metastasis | 2-year
  the number of patients with lymph node metastasis
distant metastasis | 2-year
  the number of patients with thyroid cancer metastasizing to distant tissues or organs
New thyroid cancer | 2-year
  the number of patients with new recurrent malignant thyroid tumor in other area of thyroid gland
Disease progression | 2-year
  the number of patients with local tumor progression, lymph node metastasis, new cancers or lymph node metastasis.

SECONDARY OUTCOMES:
complication rate | 2-year
  complication rate encouned during or after procedures
blood loss | 2-year
  the volume of blood loss during procedures
free thyroxine | 2-year
  change of free thyroxine concentration
free triiodothyronine | 2-year
  change of free triiodothyronine concentration
thyroid-stimulating hormone | 2-year
  change of thyroid-stimulating hormone concentration

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zheng L, Dou JP, Han ZY, Liu FY, Yu J, Cheng ZG, Yu XL, Wang H, Cong ZB, Wang SR, Yu MA, Xu ZF, Che Y, Nan B, Liu C, Hao Y, Wang X, Liu Y, Zhou Y, Liang P. Microwave Ablation for Papillary Thyroid Microcarcinoma with and without US-detected Capsule Invasion: A Multicenter Prospective Cohort Study. Radiology. 2023 May;307(3):e220661. doi: 10.1148/radiol.220661. Epub 2023 Mar 7. PMID 36880949